CLINICAL TRIAL: NCT07082790
Title: Determination of the Effect of Virtual Reality Glasses and Music Used During Non-Stress Testing on Fetal Well-Being and Anxiety in Pregnant Women
Brief Title: Effect of VR and Music on Fetal Well-Being and Anxiety During Nonstress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Rahime Aksoy, Research Assistant, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NST-2025
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Anxiety; Pregnancy; Randomised Controlled Trial; Music
Keywords: virtual reality; anxiety; pregnancy; nonstress test; music
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were divided into 3 groups (VR, music, and control). Randomization was performed via the 'Research Randomizer' (www.randomizer.org) website by a statistician from outside the study who had no previous contact with participants who met the inclusion criteria and agreed to participate in the study. This tool generated a total of 60 different codes and randomly distributed them to 3 groups. These numbers were then placed in a box, and women were assigned to a group according to the numbers they chose.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality Group (Experimental): Pregnant women in the VR group were given adaptive three-dimensional (3D) glasses that fit snugly on their heads to optimize image quality and provide full distance adjustment. All pregnant women in the group were allowed to wear the glasses for a few minutes before the application in order to get used to the glasses. The image to be projected on the glasses was provided by placing a smartphone compatible with the glasses on the front of the glasses. Pregnant women in the VR group were shown an image of a green landscape with a relaxing sound accompanying the 3D images. Pregnant women in the VR group were shown an image of green nature due to the proven psychologically relaxing effect of green. Since the content in question is prepared in 360 degrees, the person wearing the glasses finds herself in the virtual world and experiences the feeling of being there, no matter which direction she looks.
  Interventions: Other: Virtual Reality Intervention
- Music Group (Experimental): The music was provided to the pregnant women with wireless headphones worn over the head, an electronic acoustic device with sound-enhancing ear pads, and an adjustable headband. These headphones allowed the pregnant women to listen to music in isolation. The music played in the study was determined with the recommendation of the Research and Promotion of Turkish Music (TUMATA), which operates in Turkey and carries out treatment studies with Turkish music. Accordingly, pregnant women were made to listen to Acemashiran maqam, which is thought to have a positive effect on the uterus, the baby in the womb, and facilitate birth. According to TUMATA, Acemashiran Maqam has a fiery nature. It is a dry-hot makam. It is effective on bones and the brain. It helps balance fat in the body. It gives a sense of creativity and inspiration. Revitalizes stagnant thoughts and emotions. Facilitates childbirth in women. Helps to correct the wrong posture of the child in the womb.
  Interventions: Other: Music intervention
- Control Group (No Intervention): Pregnant women in the control group did not undergo any procedure and underwent routine Nonstress Test.

INTERVENTIONS:
Other: Music intervention — The music was provided to the pregnant women with wireless headphones worn over the head, an electronic acoustic device with sound-enhancing ear pads, and an adjustable headband. These headphones allowed the pregnant women to listen to music in isolation. The music played in the study was determined with the recommendation of the Research and Promotion of Turkish Music (TUMATA), which operates in Turkey and carries out treatment studies with Turkish music. Accordingly, pregnant women were made to listen to Acemashiran maqam, which is thought to have a positive effect on the uterus, the baby in the womb, and facilitate birth. According to TUMATA, Acemashiran Maqam has a fiery nature. It is a dry-hot makam. It is effective on bones and the brain. It helps balance fat in the body. It gives a sense of creativity and inspiration. Revitalizes stagnant thoughts and emotions. Facilitates childbirth in women. Helps to correct the wrong posture of the child in.
  Arms: Music Group
Other: Virtual Reality Intervention — Pregnant women in the VR group were given adaptive three-dimensional (3D) glasses that fit snugly on their heads to optimize image quality and provide full distance adjustment. All pregnant women in the group were allowed to wear the glasses for a few minutes before the application in order to get used to the glasses. The image to be projected on the glasses was provided by placing a smartphone compatible with the glasses on the front of the glasses. Pregnant women in the VR group were shown an image of a green landscape with a relaxing sound accompanying the 3D images. Pregnant women in the VR group were shown an image of green nature due to the proven psychologically relaxing effect of green. Since the content in question is prepared in 360 degrees, the person wearing the glasses finds herself in the virtual world and experiences the feeling of being there, no matter which direction she looks.
  Arms: Virtual reality Group

SUMMARY:
Music and virtual reality (VR) have been utilized in the medical field and are known to reduce anxiety and stress. However, a limited number of studies have investigated the effects of music and VR on women undergoing non-stress tests (NST). In this context, the present study aimed to determine the effects of music and VR on fetal movement, fetal heart rate, maternal physiological parameters, maternal satisfaction, and anxiety levels.

The study was conducted between June 2024 and February 2025 in the NST clinic of a training and research hospital in Bilecik, Turkey. Participants were divided into three groups: virtual reality, music, and control, with 20 pregnant women in each group. Data were collected using a personal information form, the State-Trait Anxiety Inventory, NST assessments, and a maternal parameter evaluation form.

The findings indicate that the use of VR and music during NST reduces anxiety levels in pregnant women, improves physiological parameters, and enhances satisfaction with the procedure. Notably, the decrease in anxiety levels and the positive changes in physiological parameters were more pronounced in the VR group.

The stress-reducing effects of distraction techniques such as VR and music may enhance placental blood flow, thereby positively influencing fetal movements and reactivity. However, further long-term studies are required to better understand how fetal activity is affected by emotional changes.

DETAILED DESCRIPTION:
Ethical principles were taken into consideration in the study. After the necessary arrangements were made in the data collection forms, the participants were given written and verbal explanations about the study, and their informed consent was obtained. Data collection forms were applied individually through face-to-face interviews with women who volunteered to participate in the study. A non-intervention midwife was responsible for performing NST for 20 minutes and assessing pregnant women's physiological parameters before and after NST. For pregnant women, the Personal Information Form was only administered before NST. SAI and TAI were performed before and after the NST procedure. One group of pregnant women in the intervention group was exposed to music, while the other group was exposed to virtual reality. The control group continued the routine practice. In addition, blood pressure and heart rate values of the pregnant women were measured and monitored by a midwife outside the study 5 minutes after the start of NST and after a 5-minute rest period after the end of NST. The NST assessments of the pregnant women in the group were evaluated by an obstetrician and gynecologist who was involved in the study but did not know which group the pregnant women were in.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 32 weeks,
* singleton pregnancy without any known fetal anomaly,
* no perinatal complications,
* age ≥ 18 years,
* nulliparous.

Exclusion Criteria:

* Significant medical (cardiac, renal or neurological diseases) or mental diseases (psychosis, neurosis, addictions, etc.),
* Diagnosed by a physician as high-risk pregnancy (pregnancy-related hypertension, pre-eclampsia, eclampsia, gestational diabetes, premature rupture of membranes, large or small for gestational age, intrauterine growth retardation, polyhydramnios, oligohydramnios, threatened preterm delivery),
* have a multiple pregnancy,
* have a fetus with an anomaly,
* have fetal distress for which the physician considers emergency intervention.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety | up to one hour
  The State Anxiety Inventory (SAI) and Trait Anxiety Inventory (TAI) were used to measure the anxiety levels of pregnant women. The scale was developed by Spielberger and colleagues, and its Turkish validity and reliability were examined by. The scale consists of 40 items, 20 in the SAI scale and 20 in the TAI scale. With the state anxiety scale, it is possible to determine how the individual feels at that moment and under those conditions, and with the trait anxiety scale, it is possible to determine how the individual feels in general. The scale is a 4-point Likert type. The scale includes items consisting of direct and inverted statements. When calculating the total score, the total weighted score of the direct statements is subtracted from the total weighted score of the inverted statements. To the result obtained, 50 is added for the state anxiety scale and 35 for the trait anxiety scale. The final score obtained shows the anxiety level of the individual.
Pregnancy Parameters Assessment Form | Five minutes before the non-stress test (NST)
  It is a form in which heart rate (diastolic blood pressure (DBP) and systolic blood pressure (SBP)) is assessed by a calibrated sphygmomanometer, is recorded before and after the NST procedure.
Pregnancy Parameters Assessment Form | Five minutes before the non-stress test (NST)
  It is a form in which pulse rate (maternal heart rate (MHR)), estimated by pulse oximetry, is recorded before and after the NST procedure.

SECONDARY OUTCOMES:
State-Trait Anxiety | up to one hour
  State Anxiety Inventory (SAI) and Trait Anxiety Inventory (TAI) were used to measure the anxiety levels of pregnant women. The scale was developed by Spielberger and colleagues, and its Turkish validity and reliability were examined by. The scale consists of 40 items, 20 in the SAI scale and 20 in the TAI scale. With the state anxiety scale, it is possible to determine how the individual feels at that moment and under those conditions, and with the trait anxiety scale, it is possible to determine how the individual feels in general. The scale is a 4-point Likert-type. The scale includes items consisting of direct and inverted statements. When calculating the total score, the total weighted score of the direct statements is subtracted from the total weighted score of the inverted statements. To the result obtained, 50 is added for the state anxiety scale and 35 for the trait anxiety scale. The final score obtained shows the anxiety level of the individual.
Pregnancy Parameters Assessment Form | five minutes after the non-stress test (NST)
  It is a form in which heart rate (diastolic blood pressure (DBP) and systolic blood pressure (SBP)) is assessed by a calibrated sphygmomanometer, is recorded before and after the NST procedure.
NST Parameters Evaluation | up to one hour
  The form was designed to evaluate NST results. The NST evaluation form included the fetal heart rate, acceleration, deceleration, and fetal movement counts, and the test result (reactive or non-reactive), which were monitored for at least 20 minutes.
Pregnancy Parameters Assessment Form | Five minutes after the non-stress test (NST)
  It is a form in which pulse rate (maternal heart rate (MHR)), estimated by pulse oximetry, is recorded before and after the NST procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rahime AKSOY BULGURCU, Principal Investigator — Bilecik Seyh Edebali Universitesi
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No